CLINICAL TRIAL: NCT06758180
Title: Comparison of the Learning Effects of Video-Assisted and Interactive Game-Based Approaches in Adult Basic Life Support Education: A Study of First and Emergency Aid Program Students
Brief Title: The Effect of Video-Assisted and Game-Based Approaches on Basic Life Support Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ABANT-HEM-RK-2024-379
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Basic Life Support; Student Education; Video-Assisted; Interactive Teaching
Keywords: basic life support; student; first and emergency aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Training Group (Active Comparator): One week after all students will have received verbal instruction on adult basic life support (BLS), students assigned to the Video Training Group will be provided with reinforcement training before the laboratory practice by watching a video on the topic of "Adult Basic Life Support." The video will be presented via projection by the researchers. This video will aim to reinforce students' knowledge of adult BLS.
  Video Training The video used for the training was titled "Basic Life Support and AED Usage - Adult (BLS)", which was prepared according to the 2021 ERC guidelines and made available on the 'Paramedic Online' YouTube channel as of May 31, 2023 (Paramedic Online, 2023). The video covered key topics within basic life support, including chest compressions, artificial respiration, and the use of an automated external defibrillator (AED).
  Interventions: Behavioral: verbal basic life support training; Behavioral: video training
- Interactive Video Game Group (Experimental): The intervention group will be called the video game group. After the students in this group are given verbal adult basic life support (BLS) training, reinforcement training will be provided with the interactive video game called "Lifesaver" before the laboratory application. The researcher will provide detailed information to the students about the purpose, content and use of the interactive video game, and then the game will be downloaded to the students from Google Play or the App Store.
  The students will play the game under the supervision of the researcher based on their individual reasoning. Since there is no Turkish language support during the game, the researchers will contribute to the reinforcement of correct understanding by providing translation support when necessary. The aim of the Lifesaver game is to reinforce the students' knowledge and skills on adult basic life support by taking the "Harry" scenario as the basis.
  Interventions: Behavioral: verbal basic life support training; Behavioral: Interactive game intervention

INTERVENTIONS:
Behavioral: verbal basic life support training — Both groups will be given verbal adult basic life support training simultaneously, on a day and time that will not conflict with the students' class schedules. The "Adult Basic Life Support Training" presentation published by the Ministry of Health in 2021 will be used in the training and will last approximately 40 minutes.
  A week after the verbal training, a basic life support application for adults will be held in the Faculty of Medicine Skills Laboratory.
Behavioral: Interactive game intervention — The interactive game group will be given reinforcement training before the laboratory application. Here, each student will play the game accompanied by a researcher.
  Lifesaver is an educational game developed by the Resuscitation Council (UK), offered in English and completely free of charge. The game can be downloaded to computers, phones or tablets from Google Play or the App Store. Lifesaver includes four different interactive video scenarios to help users develop their lifesaving skills. The "Harry" scenario to be used in this research is based on a real case. In the scenario, Harry, a high school student who has a sudden heart attack while playing football, is given heart massage, CPR and defibrillation by his friends.
  The game offers different options at each stage to improve the players' knowledge and skill levels. If a wrong choice is made, the same section is played again until the correct step is performed. The completion time of the game may vary average 15 minutes.
  Arms: Interactive Video Game Group
Behavioral: video training — One week after all students are given verbal adult basic life support training, a video titled "Adult Basic Life Support" will be shown to the students in the video training group before the laboratory application. The video will be shown by the researcher using a projector. After the video watching process is completed, each student will apply basic life support on the adult training model in turn and the applications will be evaluated individually. In the video training, the video titled "Basic Life Support and AED Use - Adult (TYD)", which was published as open access on the 'paramedic online' YouTube channel on May 31, 2023 and prepared in accordance with the 2021 ERC guideline, will be used (Paramedic online, 2023). This video covers the topics of heart massage, artificial respiration and automatic external defibrillator use within the scope of basic life support.
  Arms: Video Training Group

SUMMARY:
Adult Basic Life Support (BLS) is a critical skill in emergency situations. Teaching this skill effectively to students in first aid and emergency aid programs is essential for imparting both theoretical knowledge and practical competencies. Educational methods have a direct impact on students' knowledge levels and skill acquisition. In addition to traditional teaching methods, advancements in educational technology have introduced innovative approaches such as interactive video games into this field. This study compares the effects of two different instructional methods-video-assisted education and interactive video game-supported education-on students' learning outcomes and practical performance in adult BLS training.

DETAILED DESCRIPTION:
**Basic Life Support (BLS)** refers to non-pharmacological interventions performed to sustain life by pumping blood from the heart through external chest compressions and delivering oxygen to the lungs via artificial respiration for individuals showing no signs of life (chest movement, coughing, any bodily movement, or pulse). In cases where critical risks persist in the circulatory and respiratory systems, if BLS interventions are not promptly initiated, brain damage can occur within 4-6 minutes after the cessation of respiration and circulation. If the oxygen deprivation to brain tissue exceeds 10 minutes, irreversible brain damage ensues.Therefore, considering the critical importance of BLS in both prehospital and in-hospital cardiac arrest situations, BLS training is incorporated as a mandatory course in the curriculum for students in First and Emergency Aid programs.

Despite the transformative role of digital technologies in education in recent years, globally, BLS training is predominantly conducted using traditional methods. In the traditional approach, the instructor initially provides theoretical knowledge on BLS and then conducts practical skill training using CPR mannequins. At the end of the training, students practice what they have learned on the mannequin under the instructor's supervision. However, research indicates that, despite its widespread use, the traditional method alone is insufficient and that knowledge and skills acquired through this approach may fade over time. The primary limitations of the traditional method include large class sizes, insufficient instructor numbers, time constraints, and the limited opportunity for each student to practice adequately.

On the other hand, various studies emphasize the importance of traditional education and suggest that its effectiveness can be enhanced, and the retention of skills prolonged when supplemented with alternative methods. For instance, a study by Castillo et al. (2020) highlighted that hybrid approaches combining traditional BLS training with other instructional methods improved knowledge retention. Therefore, it is recommended that traditional methods be supported by evidence-based new approaches to enhance educational efficiency. Among these methods, video-assisted training, when combined with face-to-face theoretical education, has been shown to improve students' knowledge and skill levels in BLS. However, research on this subject remains limited, and the ideal methodology for teaching correct intervention knowledge and skills in cardiac arrest and ensuring their retention has yet to be determined. To achieve the goal of delivering high-quality resuscitation, further exploration of new methodologies and technologies is needed.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of the first and emergency aid program
* Not having received any previous training on basic life support
* Understanding and speaking Turkish
* Voluntarily accepting to participate in the research

Exclusion Criteria:

* Being on leave of absence, being on sick leave, being absent during the implementation process of the research,
* Being a foreign national,
* Not accepting to participate in the research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
knowledge level | before oral training, 1 week after oral training, 2 months after oral training
  The knowledge level measurement will be made using the "Basic Life Support Knowledge Level Assessment Form". This form was prepared to evaluate the participants' theoretical knowledge levels about adult basic life support (BLS) and consists of 15 multiple-choice questions.
  Measurement Process:
  1. Pre-Test: Before participating in the study, students in both groups will be asked to fill out the form to measure their knowledge levels before the training is given.
  2. Post-Test:1 week after the verbal training, all students will be asked to fill out the form to re-evaluate their knowledge levels.
  3. Follow-up test: Approximately 2 months after the training students in both groups will be asked to fill out the form to re-evaluate their knowledge levels.
  Form Content: The form was created by the researchers through a literature review. All measurements are planned to be carried out face-to-face in an average of 15 minutes.
skill level | during the laboratory practice to be held 1 week after the oral training, during the laboratory practice to be held 2 months after the oral training
  In this study, students' basic life support (BLS) skill levels will be measured twice using the "Basic Life Support Skills Assessment Form".
  1. Interactive Video Game Group:
     After playing the interactive video game called Lifesaver, students will individually practice BLS on a model in the Medical Faculty Skills Laboratory.
     Researchers will observe students' performances during the application and evaluate each item on the form as "Sufficient" (2 points), "Needs Improvement" (1 point) or "Inadequate" (0 points).
     The scores received by each student in the group will be used to analyze the effectiveness of this method.
  2. Video Training Group:
  After watching the video training on BLS, students will individually practice BLS on a model in the skill laboratory.
  Their performances will again be evaluated according to the same criteria using the "Basic Life Support Skills Assessment Form".

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Can Cicek, Assoc Prof, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No